CLINICAL TRIAL: NCT07033975
Title: A Flavonoid-enriched Mediterranean Diet for Multiple Sclerosis
Brief Title: A Specialized Diet for Multiple Sclerosis
Acronym: FLAMEMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jerome J. A. Hendriks (Other)
Collaborators: Revalidatie & MS Centrum Overpelt (Other)
Responsible Party: Sponsor-Investigator, Jerome J. A. Hendriks, Prof. Dr. Jerome J.A. Hendriks, Hasselt University
Organization: Hasselt University (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: B1152023000003
Record Dates: First submitted 2025-04-24; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Flavonoid-enriched Mediterranean Diet (Experimental)
  Interventions: Other: Flavonoid-enriched Mediterranean Diet

INTERVENTIONS:
Other: Flavonoid-enriched Mediterranean Diet — A set of dietary guidelines describing an adjusted Mediterranean diet focusing on the intake of flavonoid-rich products.

SUMMARY:
This study examines the impact of a Mediterranean diet on individuals with multiple sclerosis (MS). MS is a multifactorial disease in which environmental factors, such as nutrition, can influence disease progression. Therefore, this study aims to investigate whether a healthier dietary pattern, specifically a flavonoid-rich Mediterranean diet, can affect disease parameters.

ELIGIBILITY:
Inclusion Criteria:

* Expanded Disability Status Scale (EDSS): 0-6

Exclusion Criteria:

* Diagnosed digestive pathology

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-04 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Microbiota changes | Three timepoints, before start of the strict diet (day 14), after the strict diet (day 31), and after the follow-up period of three months (day 122).
  Microbiota sequencing on fecal samples to identify the different bacterial strains that are present.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasselt University, Diepenbeek, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: Undecided